CLINICAL TRIAL: NCT05601024
Title: The Effect of Laughter Therapy on Self-Esteem and Quality of Life in Patients With Stoma:Randomized Controlled Trial
Brief Title: The Effect of Laughter Therapy on Self-Esteem and Quality of Life in Patients With Stoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hatice Merve Alptekin, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-74555795-050.01.04-97020
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Stoma Colostomy; Stoma Ileostomy
Keywords: Laughter Therapy; Quality of Life; Self Esteem; Stoma
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 1. After obtaining permission from the participants, patients will be called by phone and questions will be asked about Rosenberg Self-Esteem Scale, sociodemographic characteristics, City of Hope Quality of Life Ostomy.
  2. Participants in this group will receive a 4 week of laughter therapy. Laughter therapy will be conducted on whatsapp.
  3. After laughter therapy (after 1 month): Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.
  4. After 3 month: Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.
  Interventions: Behavioral: Laughter Therapy
- Control Group (No Intervention): 1. After obtaining permission from the participants, patients will be called by phone and questions will be asked about Rosenberg Self-Esteem Scale, sociodemographic characteristics, City of Hope Quality of Life Ostomy.
  2. After 2 weeks: Patients will be called by phone and asked if they have any complaints about their disease.
  3. After 1 month: Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.
  4. After 3 month: Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.

INTERVENTIONS:
Behavioral: Laughter Therapy — The first component of intervention is the laughter therapy that is a combination of warm up exercise, deep breathing exercises, childlike playfulness and laughter exercises. Participants will do laughter therapy with whatsapp group call. Each group will consist of at least 5 people. Each session of laughter therapy will be offered one a weekly and 30-40 minutes each time.
  Arms: Experimental Group

SUMMARY:
Stoma is a surgical intervention to ensure that body wastes are removed differently from the normal physiological opening. The stoma patient has to cope with complex emotional, social and physical problems associated with this change. Physical health problems (such as stoma), change in body image and negative emotions affect self-esteem and quality of life. Laughing provides mental and physical relaxation with the release of endorphins. Therefore, laughter therapy has an important contribution to increase the well-being of patients.This study was planned as a randomized controlled experimental study to evaluate the effect of laughter therapy on self-esteem and quality of life in patients with stoma.

DETAILED DESCRIPTION:
The total number of individuals with a stoma is thought to be between 725,000 and 1 million (Faqs, 2020). Stoma can cause many physical, social, cognitive and emotional problems in an individual's life. These problems can negatively affect the quality of life of patients with stoma (Karadag et al. 2011).

Self-esteem is an individual's positive or negative evaluation of himself/herself (Ayaz, 2008). This evaluation stems not from the individual's need to feel perfect, but from the need to accept himself and be accepted by others. Physical health problems, changes in body image and negative emotions affect self-esteem.

Laughter is generally considered to be a visual expression of happiness or a feeling of joy, and it occurs with stimuli such as hearing a joke or being tickled. Neurophysiology has shown that laughter is associated with the activation of the lower middle frontal lobe cortex, which produces endorphins (Satish 2012). Laughing provides mental and physical relaxation with the release of endorphins (Farifteh et al. 2014).

Psychological benefits of laughing;

* Decreases symptoms of depression, anxiety and stress level.
* Increases self-confidence, hope, energy and strength.
* Increases memory, creative thinking and problem solving ability.
* Increases interpersonal relationship and social interaction.
* Collaboration enhances group identity and solidarity.
* Strengthens the relationship between the health personnel and the patient.
* Provides psychological well-being.
* Increases joy and it's mostly contagious (Ripoll and Casado 2010).

It was found to increase optimism and self-esteem in a study of menopausal women (Cha et al. 2013). As a result of Cho and Oh's (2011) study, it was stated that laughter therapy can be an effective nursing intervention applied to increase the quality of life and recovery in individuals with breast cancer. Although laughing therapy was applied in different patient groups and its positive effects were proven, a study on patients who had undergone surgical intervention could not be reached. This study was planned as a randomized controlled experimental study to evaluate the effect of laughter therapy on self-esteem and quality of life in patients with stoma.

Study Population and Sampling: In the study, in calculating the sample size to be used to measure the effect of laughter therapy on self-esteem and quality of life in patients with stoma, the d value was determined as d = 0.66, α = 0.05 (margin of error), 1-β = 0.95 (power) in the light of academic studies. With the help of the G-power (version 3.1) package program, the number of samples to be included in the study was calculated as 68 people (Yoshikawa et al. 2019). Considering a possible 10% loss in the study, it was decided to include a total of 74 participants, 37 participants in each group.

Randomization: The research was conducted as an open-label, blinded, randomized and controlled experimental study. A simple computer-assisted randomization method was used to distribute the groups homogeneously.

For this purpose, 74 sets were created using the functions available on the "https://www.random.org/integer-sets" website. In each of these sets, there were a total of 8 participants: 4 participants from the experimental group and 4 participants from the control group. The 74 sets created as the next process were shown with 1 number each. "RANDBETWEEN" function was used in Excel. Thus, 10 numbers between 1 and 74 were generated and 10 sets to be used in randomization were randomly determined. 72 patients were randomized in the first 9 sets and 2 patients in the 10th set.

Data Collection Method: Data will be collected by the researcher by calling the participants by phone. WhatsApp video chat method will be applied for the individuals in the experimental group.

Data Collection Tools:

1. Personal information form (sociodemographic characteristics): With this form, which was prepared by the researcher in line with the literature, it is planned to obtain information about the sociodemographic characteristics (gender, age, occupation, etc.) and stoma (diagnosis, stoma type, etc.) of the participants.
2. Rosenberg Self-Esteem Scale: Rosenberg Self-Esteem Scale was developed by Morris Rosenberg in 1965. In 1985, The validity and reliability study of the scale, which was translated into Turkish by Dr. Füsun Çetin Çuhadaroğlu, was also conducted by Çuhadaroğlu (Çuhadaroğlu, 1986). This scale consists of 10 questions that measure self-esteem. IThe highest score that can be obtained from the scale is 6.
3. City of Hope Quality of Life Ostomy: The scale was developed by the Hope Center Pain and Palliative Care Research Center in 1995 to evaluate the quality of life of cancer patients. It is a 43-item Likert-type scale revised for individuals with ostomy. The Turkish adaptation and validity-reliability study of the scale was carried out by Erol and Vural (2012).

Intervention:

The first component of intervention is the laughter therapy that is a combination of warm up exercise, deep breathing exercises, childlike playfulness and laughter exercises.

Hand clapping and warm-up exercises: Hands are kept parallel to each other and clapped so that the fingertips touch each other. In order to synchronize the group and increase the energy level of the group, rhythms such as ho-ho, ha-ha-ha are usually added to the clapping.

Deep breathing exercises: Deep breathing exercises are exercises for filling and emptying the lungs, providing physical and mental relaxation. It is applied by breathing through the nose and exhaling slowly through the mouth.

Childlike acting: One of the purposes of the laughing exercises is that childlike acting comes to life in the mind and helps to laugh. During this exercise, songs can be sung, games can be played, and laughing can be helped with music.

Laughter exercises: yogic laugh exercises (Lion laugh), cheerful laugh exercises (milkshake, hot soup laugh) and physical laughter exercises.

Participants will do laughter therapy with whatsapp group call. It is important for participants to share their images and voices in order to make eye contact and hear the sounds of laughter. Each group will consist of at least 5 people. Each session of laughter therapy will be offered one a weekly and 30-40 minutes each time.

Experimental Group

* After obtaining permission from the participants, patients will be called by phone and questions will be asked about Rosenberg Self-Esteem Scale, sociodemographic characteristics, City of Hope Quality of Life Ostomy.
* Participants in this group will receive a 4 week of laughter therapy. Laughter therapy will be conducted on whatsapp.
* After laughter therapy (after 1 month): Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.
* After 3 month: Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.

Control Group

* After obtaining permission from the participants, patients will be called by phone and questions will be asked about Rosenberg Self-Esteem Scale, sociodemographic characteristics, City of Hope Quality of Life Ostomy.
* After 2 weeks: Patients will be called by phone and asked if they have any complaints about their disease.
* After 1 month: Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.
* After 3 month: Patients will be called again by phone to ask questions about the Rosenberg Self-Esteem Scale and City of Hope Quality of Life Ostomy.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Being able to understand and speak Turkish,
* Stoma has been opened at least 6 months ago,
* To have completed oncological treatments,
* Having a smart phone or computer,
* Being able to use a smart phone or computer,
* Having internet,
* Being able to use Whatsapp video calling program,
* Agreeing to participate in the research.

Exclusion Criteria:

* Hernia, prolapse of stoma complications or glaucoma disease,
* Presence of hypertension and heart disease,
* Abdominal surgery in the last 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
City of Hope Quality of Life Ostomy | Change from baseline to 1 months
  This scale, which evaluates the quality of life, consists of 43 items. In this scale, quality of life items are grouped into four sub-dimensions: physical well-being (1-11 items), psychological well-being (12-24 items), social anxiety (25-36 items) and spiritual well-being (37-43 items).
Rosenberg Self-Esteem Scale | Change from baseline to 1 months
  This scale consists of 10 questions that measure self-esteem. If the total score from 10 questions is 0-1, it indicates high self-esteem, 2-4 indicates medium, and 5-6 indicates low self-esteem. The highest score that can be obtained from the scale is 6

SECONDARY OUTCOMES:
City of Hope Quality of Life Ostomy | Change from baseline to 3 months
  Changes in patients' longer-term quality of life will be assessed after laughter therapy.
Rosenberg Self-Esteem Scale | Change from baseline to 3 months
  Changes in patients' longer-term self-esteem will be assessed after laughter therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Akyüz, Associate Professor, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Hatice Merve Alptekin, Istanbul, Sisli, Turkey (Türkiye)

REFERENCES:
- [Background] Karadag A, Ozturk D, Celik B. Adaptation of the ostomy adjustment inventory into Turkish Language. Turk J Colorectal Dis. 2011;21:173-181.
- [Background] Ayaz S. Body image and self-esteem in patients with stoma: Review. Turkiye Klinikleri J Med Sci. 2008; 28(2):154-159.
- [Background] Satish PD. Laughter therapy. Journal of Pharmaceutical and Scientific Innovation. 2012;1(3):23-4.
- [Background] Farifteh S, Mohammadi-Aria A, Kiamanesh A, Mofid B. The Impact of Laughter Yoga on the Stress of Cancer Patients before Chemotherapy. Iran J Cancer Prev. 2014 Fall;7(4):179-83. PMID 25628838
- [Background] Ripoll RM, Casado IQ. Laughter and positive therapies: modern approach and practical use in medicine. Rev Psiquiatr Salud Ment. 2010 Jan;3(1):27-34. doi: 10.1016/S1888-9891(10)70006-9. Epub 2010 Apr 14. English, Spanish. PMID 23017490
- [Background] Cha MY, Na YK, Hong HS. An Effect of Optimism, Self-esteem and Depression on Laughter Therapy of Menopausal Women. Korean J Women Health Nurs. 2012 Dec;18(4):248-256. doi: 10.4069/kjwhn.2012.18.4.248. Epub 2012 Dec 31. PMID 37697500
- [Background] Cho EA, Oh HE. [Effects of laughter therapy on depression, quality of life, resilience and immune responses in breast cancer survivors]. J Korean Acad Nurs. 2011 Jun;41(3):285-93. doi: 10.4040/jkan.2011.41.3.285. Korean. PMID 21804337
- [Background] Yoshikawa Y, Ohmaki E, Kawahata H, Maekawa Y, Ogihara T, Morishita R, Aoki M. Beneficial effect of laughter therapy on physiological and psychological function in elders. Nurs Open. 2018 Jul 18;6(1):93-99. doi: 10.1002/nop2.190. eCollection 2019 Jan. PMID 30534398
- [Background] Çuhadaroğlu F. (1986).Adolesanlarda Benlik Saygısı, Hacettepe Üniversitesi Tıp Fakültesi, Psikiyatri Anabilim Dalı, Uzmanlık Tezi, Ankara
- [Background] Erol F, Vural F. Validity and reliability of the city of hope quality of life ostomy -scale forthe Turkish patients with ostomy. Hemşirelikte Araştırma Geliştirme Dergisi. 2012;3.
- See also: Living with an Ostomy: FAQS — https://www.ostomy.org/living-with-an-ostomy/